CLINICAL TRIAL: NCT04256122
Title: Expression of Markers Related to Mitochondrial Functionality in Carcinoma of the Urinary Bladder: Comparative Retrospective Analysis Between Recurrent Tumors ("Non-responders") and Non-recurrent Tumors ("Responders") After Intravesical Treatment With Chemotherapy or Immunotherapy
Acronym: MITOMARKER-MIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Clinical Research, Istituto Clinico Humanitas
Other Study IDs: 1191
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responder patients: Patients with NMIBC at first diagnosis, pTa/pT1 (primary tumors) treated with MMC or BCG after TURBT will be selected from the institutional patient registry.
  * Patient treated with adjuvant MMC or BCG that did not experience recurrence for at least 42 months after TURBT
  * Patients are tumor-free at the moment of the analysis
  Interventions: Other: No intervantion on patients. retrospective study is performed on paraffin embedded tumor tissue specimens routinely collected during TURBT.
- Non responder patients: Patients with NMIBC at first diagnosis, pTa/pT1 (primary tumors) treated with MMC or BCG after TURBT will be selected from the institutional patient registry.
  o Patient treated with adjuvant MMC or BCG that experienced recurrence in the first 24 months after TURBT.
  Interventions: Other: No intervantion on patients. retrospective study is performed on paraffin embedded tumor tissue specimens routinely collected during TURBT.

INTERVENTIONS:
Other: No intervantion on patients. retrospective study is performed on paraffin embedded tumor tissue specimens routinely collected during TURBT. — evaluate an immunophenotypical profile related to mitochondrial functions in tumors responders vs non-responder to intravescical chemotherapy or immunotherapy. Verify the possible prognostic differences in clinical behavior between the two populations.

SUMMARY:
Retrospective monocentric study evaluating different immunohistochemical phenotypes related to mitochondrial functions with treatment outcomes

DETAILED DESCRIPTION:
About 80% of newly diagnosed patients have non-muscle-invasive bladder cancer (NMIBC), including papillary lesions confined to the urothelium (stage Ta) or invading the lamina propria (stage T1), and carcinoma in situ (CIS). These tumors show low progression rates, but high recurrence. In particular, patients with multifocal high-grade urothelial carcinoma have a high risk of both recurrence (∼70% after 1 yr) and progression (5% after 1 yr). Initial NMIBC management is a transurethral resection of bladder tumor (TURBT), followed by adjuvant intravesical treatment with the chemotherapeutic agent Mitomycin C (MMC) or the immunotherapy Bacillus Calmette-Guérin (BCG). However, these therapies lead to variable clinical responses and patients recur shortly after surgery. Despite both therapies have been used for decades in the treatment of NMIBC, at the moment it is not possible to predict after initial staging which patients will benefit from them since neither resistance mechanisms nor genetic markers associated to relapse have been identified yet.

In a preliminary analysis, the invesitigators found that low expression of several proteins involved in mitochondrial functions correlate with a worst prognosis in bladder cancer patients. The aim of this study is to detect markers of mitochondrial dysfunction by immunohistochemistry in recurrent tumors ("non-responders") and non-recurrent tumors ("responders") after intravesical treatment with chemotherapy or immunotherapy, and determine the prognostic relevance of these different markers.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age at diagnosis
* Histologically confirmed NMIBC urothelial carcinoma of the urinary bladder (pTa, pT1, CIS)
* Primary NMIBC or not treated secondary NMIBC, after a primary non-invasive malignancy
* Patients underwent TURBT for NMIBC at Humanitas between 2000 and 2019
* Patients that received intravesical instillations with either MMC or BCG after TURBT at Humanitas between 2000 and 2019
* Written informed consent to research purpose
* For non-recurrent tumors ("responders"):

  * Patient treated with adjuvant MMC or BCG that did not experience recurrence for at least 42 months after TURBT
  * Patients are tumor-free at the moment of the analysis
* For recurrent tumors ("non-responders"):

  * Patient treated with adjuvant MMC or BCG that experienced recurrence in the first 24 months after TURBT.

Exclusion Criteria:

* Previous malignancies other that bladder cancer
* Patients with a history of treated bladder cancer recurrences

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with NMIBC at first diagnosis, pTa/pT1 (primary tumors) treated with MMC or BCG after TURBT will be selected from the institutional patient registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemestry analysis of biomarkers | 1 year
  perform an immunophenotypical analysis to assess the expression of key proteins involved in mitochondrial functionality in recurrent tumors ("non-responders") and non-recurrent tumors ("responders") after intravesical treatment with chemotherapy or immunotherapy.

SECONDARY OUTCOMES:
Correlation of biomarker expression with outcome | 1 year
  • To correlate the resulting phenotype with clinical/pathological response to adjuvant treatments (time to recurrence and presence of recurrence).

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas reseach hospital (ICH), Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Research outcome

REFERENCES:
- [Derived] Oresta B, Pozzi C, Braga D, Hurle R, Lazzeri M, Colombo P, Frego N, Erreni M, Faccani C, Elefante G, Barcella M, Guazzoni G, Rescigno M. Mitochondrial metabolic reprogramming controls the induction of immunogenic cell death and efficacy of chemotherapy in bladder cancer. Sci Transl Med. 2021 Jan 6;13(575):eaba6110. doi: 10.1126/scitranslmed.aba6110. PMID 33408185